CLINICAL TRIAL: NCT00093080
Title: A Phase II Study of AP23573, An mTOR Inhibitor, in Patients With Advanced Sarcoma
Brief Title: Study of AP23573/MK-8669 (Ridaforolimus), A Mammalian Target of Rapamycin (mTOR) Inhibitor, in Participants With Advanced Sarcoma (MK-8669-018 AM1)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-018; AP23573-04-202 (Other: Ariad Pharmaceuticals, Inc.); 2004-002231-92 (EudraCT Number)
Record Dates: First submitted 2004-09-30; First posted 2004-10-04 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Leiomyosarcoma; Liposarcoma; Osteosarcoma; Sarcoma, Soft Tissue; Metastases
Keywords: Metastatic and/or unresectable soft tissue or
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Osteosarcoma; Sarcoma; Neoplasm Metastasis | interventions — ridaforolimus

ARMS (1):
- Ridaforolimus (Experimental): 12.5 mg of ridaforolimus is given intravenously over 30 minutes once daily for 5 days, every 2 weeks
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — 12.5 mg of ridaforolimus is given intravenously over 30 minutes once daily for 5 days, every 2 weeks
  Other Names: deforolimus (until May 2009); AP23573; MK-8669

SUMMARY:
The purpose of this study is to assess the efficacy of ridaforolimus when administered once daily for 5 consecutive days (QDx5) every two weeks in participants with advanced sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥15 years of age with metastatic and/or unresectable sarcomas of the following histological subgroups: Bone sarcomas, such as osteosarcoma and Ewings sarcoma; Leiomyosarcoma; Liposarcomas; Any other soft tissue sarcoma except gastrointestinal stromal tumors (GIST). Patients with well-differentiated liposarcoma or desmoid tumors must have demonstrated progressive disease within the previous 6 months
* Presence of at least one measurable lesion that: Can be accurately measured in at least one dimension with longest diameter ≥20 mm using conventional techniques or ≥10 mm with spiral computerized tomography (CT) scan (or otherwise at least twice the reconstruction interval for CT or magnetic resonance imaging [MRI] scans)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Minimum life expectancy of 3 months
* Adequate renal and hepatic function, as specified in the protocol
* Adequate bone marrow function, as specified in the protocol
* Serum cholesterol <350 mg/dL and triglycerides < 400 mg/dL
* Male and female patients who are not surgically sterile or postmenopausal must agree to use reliable methods of birth control for the duration of the study until 30 days after the last dose of study drug
* Able to understand and give written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Presence of brain metastases
* Prior therapy with rapamycin, rapamycin analogues or tacrolimus
* Prior anticancer treatment (chemotherapy, radiotherapy, hormonal, immunotherapy, biological response modifiers, signal transduction inhibitors, etc) within 4 weeks prior to the first dose of ridaforolimus
* Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ grade 1 by National Cancer Institute (NCI) toxicity criteria)
* Another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinoma in situ)
* Known or suspected hypersensitivity to drugs formulated with polysorbate 80 (Tween) or any other excipient contained in the study drug
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
* Significant uncontrolled cardiovascular disease
* Active infection requiring systemic therapy
* Known human immunodeficiency virus (HIV) infection
* Treatment with any investigational agent within 4 weeks prior to the first dose of ridaforolimus
* Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for 2 weeks prior to first planned dose of study drug
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of ridaforolimus
* Presence of any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluating the safety of the study drug

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Clinical Benefit Response (CBR) Using Response Criteria in Solid Tumors (RECIST) | Day 1 up to 4 years or discontinuation from study

SECONDARY OUTCOMES:
Time to Tumor Progression | Day 1 up to the first observation of disease progression, death, or the date of the last evaluation of response (up to 4 years)
Progression Free Survival | Day 1 to the first observation of disease progression, death, or the date of the last evaluation of response (up to 4 years)
Overall Survival | Day 1 to the date of death, or the date of last contact (up to 4 years)
Duration of Response | Day 1 up to the first observation of disease progression, death, or the date of the last evaluation of response (up to 4 years)
Number of participants experiencing adverse events | From first dose up to 30 days after last dose (up to 1 year)
Number of participants who discontinued study drug due to adverse events | From first dose up to the last dose (up to 1 year)
Mean ridaforolimus blood levels within 5 minutes post intravenous infusion | Day 1 and Day 5 of Cycle 1

REFERENCES:
- [Result] Chawla SP, Staddon AP, Baker LH, Schuetze SM, Tolcher AW, D'Amato GZ, Blay JY, Mita MM, Sankhala KK, Berk L, Rivera VM, Clackson T, Loewy JW, Haluska FG, Demetri GD. Phase II study of the mammalian target of rapamycin inhibitor ridaforolimus in patients with advanced bone and soft tissue sarcomas. J Clin Oncol. 2012 Jan 1;30(1):78-84. doi: 10.1200/JCO.2011.35.6329. Epub 2011 Nov 7. PMID 22067397